CLINICAL TRIAL: NCT02136290
Title: Randomized Clinical Trial of Portion-Controlled Prepackaged Foods to Promote Weight Loss - CHOICES Study.
Brief Title: Prepackaged Foods to Promote Weight Loss
Acronym: CHOICES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Cheryl Rock, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 140047; Nestle (Registry Identifier: Nestle)
Record Dates: First submitted 2014-01-08; First posted 2014-05-13 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Overweight; Obese
Keywords: Weight loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Other): Weight loss counseling
  Interventions: Behavioral: Usual Care
- Prepackaged meal (Experimental): Prepackaged meals
  Interventions: Behavioral: Prepackaged meals

INTERVENTIONS:
Behavioral: Prepackaged meals — Portion-controlled prepackaged meals
  Arms: Prepackaged meal
Behavioral: Usual Care — Usual care dietary counseling
  Arms: Usual Care

SUMMARY:
The primary goal of this clinical trial is to examine whether provision of portion-controlled prepackaged foods in the context of a reduced-energy diet prescription and counseling is associated with a greater degree of weight loss at three months in overweight or obese men and women, compared to usual care or control conditions in which the prescribed reduced-energy diet is to be consumed via self-selected foods. The effect on body weight and recognized indicators of disease risk, diet quality and cardiopulmonary fitness, as well as meal satiety and satisfaction, will also be examined. Participants are 184 overweight or obese men and women in San Diego area who will be randomly assigned to usual care or control conditions.

DETAILED DESCRIPTION:
The first study aim is (1) to test, in a randomized controlled trial, whether provision of portion-controlled prepackaged lunch and dinner entrees in the context of a reduced-energy diet prescription and counseling is associated with a greater degree of weight loss at 12 weeks in overweight or obese men and women, compared to usual care or control conditions in which the prescribed reduced-energy diet is to be consumed via self-selected foods. This study utilizes a randomized study design with participants assigned to the prepackaged food intervention arms or a usual care control group. The second study aim is (2) to describe the effect of participation in the prepackaged food arms (versus control conditions) on circulating lipids (fasting total plasma cholesterol and triglycerides, low-density lipoprotein [LDL] cholesterol, and high-density lipoprotein [HDL] cholesterol), carotenoids (a biomarker of vegetable and fruit intake), C-reactive protein, and cardiopulmonary fitness.

Secondary aims of this study are (3) to describe the association between prepackaged food consumption on meal satiety, eating attitudes and behavior, and meal satisfaction. The hypothesis to be tested is that eating a reduced-energy diet that incorporates unit-defined, prepackaged foods is associated with meal satiety and satisfaction that is superior to a diet based on self-selected foods.

As an exploratory aim, we also will examine whether there is a differential response to different dietary macronutrient composition in the prepackaged food items used in the structured meal plan in intervention participants. Lean Cuisine meal products will be offered to participants assigned to one intervention group, and only Lean Cuisine items with protein contributing >25% energy will be offered to participants in the other intervention group.

Notably, the results of this study may contribute valuable data to the scientific knowledge base regarding the various aspects of diet and diet composition that may promote more successful weight loss. How diet can be best modified to promote weight loss is an important issue currently being considered and debated among clinical and community-based behavioral and nutritional scientists, and the optimal composition for weight loss diets has not been established (IOM 2002). Adherence to any dietary regimen and energy imbalance is a central determinant of successful weight loss, and evidence-based approaches that may promote better adherence with less deprivation and more meal satisfaction could help public health and clinical efforts to reduce the high prevalence of overweight and obesity in the U.S. today.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese men and women
* Aged 25-65 years
* initial BMI >27.0 kg/m2 and < 40 kg/m2
* no eating disorders, food allergies or intolerances
* no history of bariatric surgery
* willing and able to participate in clinic visits and study interactions at specified intervals
* maintain contact with the investigators for at least three months
* willing to allow blood collections
* capable of performing a simple test for assessing cardiopulmonary fitness

Exclusion Criteria:

* inability to participate in physical activity because of co-morbidity or disability (e.g., severe arthritic conditions);
* a history or presence of a comorbid disease for which diet modification and increased physical activity may be contraindicated or complicated;
* self-reported pregnancy or breastfeeding or planning a pregnancy within the next two years;
* currently actively involved in another diet intervention study or organized weight loss program;
* a history or presence of a significant psychiatric disorder or any other condition that, in the investigator's judgment, would interfere with participation in the trial.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Weight loss | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L Rock, PhD, RD, Principal Investigator — UC San Diego Moores Cancer Center
Locations (2):
- United States (2):
  - University of California, San Diego, Moores Cancer Center, La Jolla, California
  - University of California, San Diego, La Jolla, California